CLINICAL TRIAL: NCT00396136
Title: Corox OTW Steroid LV Lead Monitoring
Brief Title: COSMO Post Approval Registry: Corox OTW Steroid LV Lead Monitoring
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20061550
Record Dates: First submitted 2006-11-01; First posted 2006-11-06 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-04

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure; Cardiac Resynchronization Therapy; Left Ventricular Lead
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Device: Corox OTW Steroid Left Ventricular Lead — This is a registry: no study required interventions necessary.

SUMMARY:
The objective of this post approval registry is to confirm the long-term safety and effectiveness of the Corox Over-the-wire (OTW) Steroid Left Ventricular (LV) lead as used in conjunction with a BIOTRONK cardiac resynchronization therapy defibrillator (CRT-D). The Corox OTW Steroid LV Lead is capable of providing permanent pacing therapy to the left ventricle in a CRT-D system. The following are the specific objectives to be evaluated during this post-approval registry:

* Long-term effectiveness of the COROX OTW Steroid in providing biventricular pacing
* Safety of the COROX OTW Steroid LV pacing lead

DETAILED DESCRIPTION:
This post approval registry enrolled 221 patients from 34 centers. The collection of registry data continued for three years for each enrolled subject. Potential patients were screened by the enrolling physician according to the detailed inclusion and exclusion criteria below.

The specific required visits for this registry are: Enrollment, Three-month, Six month, One-year, Routine Follow-Ups (every subsequent 6 months), Interim follow-ups for Corox OTW Steroid LV lead related visits, and Out of Service visit. Data will be collected at each patient follow-up. The programmed pacing parameters, LV pacing impedance, and LV pacing threshold measurement at 0.5ms pulse width will be obtained. The programming parameters will be set to best suit each patient. If adequate system function, including effective CRT, cannot be obtained, the patient should not be selected for the registry.

ELIGIBILITY:
Inclusion Criteria:

* Successfully implanted BIOTRONIK CRT-D system, including the Corox OTW Steroid LV Lead, from 1-30 days prior to enrollment
* Able to understand the nature of the registry and give informed consent
* Available for follow-up visits on a regular basis at the investigational site
* Age greater than or equal to 18 years

Exclusion Criteria:

* Enrolled in another cardiovascular or pharmacological clinical investigation
* Planned cardiac surgical procedures or interventional measures within the next 6 months
* Expected to receive a heart transplant within 6 months
* Life expectancy less than 6 months
* Presence of another life-threatening, underlying illness separate from their cardiac disorder
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2006-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katerina de Metz, Study Director — Biotronik, Inc.
Locations (1):
- Biotronik, Lake Oswego, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Corox OTW Unipolar Lead: Study Participants followed for three years post implant.
Period: Overall Study
Arm/Group | Corox OTW Unipolar Lead
Started | 221
Completed | 96
Not Completed | 125
Not completed — Death | 43
Not completed — Withdrawal by Subject | 59
Not completed — Lost to Follow-up | 15
Not completed — Study device explanted | 8

BASELINE CHARACTERISTICS:
Arm/Group | Corox OTW Unipolar Lead
Number analyzed (Participants) | 221
Age Continuous [Mean (Standard Deviation); unit: years] | 67.3 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 168
Region of Enrollment [Number; unit: participants]
  United States | 221

OUTCOME MEASURES:

1. Primary Outcome: Long-term Effectiveness of the COROX Over-the-wire (OTW) Steroid in Providing Biventricular Pacing
Description: Evaluate threshold voltage of the COROX OTW Unipolar Lead.
Time Frame: All follow-ups for 3 years post implant
Population: All study participants.
Measure: Mean (Standard Deviation); unit: Threshold Voltage
Units Other Than Participants: LV Lead Threshold Tests
Arm/Group | Corox OTW Unipolar Lead
Number analyzed (Participants) | 221
Number analyzed (LV Lead Threshold Tests) | 1130
Threshold Voltage | 1.3 (1.1)

2. Primary Outcome: Safety of the COROX OTW Steroid LV Pacing Lead
Description: Number of participants with LV lead related adverse events requiring additional invasive intervention to resolve.
Time Frame: 3 years post implant
Population: All study participants.
Measure: Number; unit: participants
Arm/Group | Corox OTW Unipolar Lead
Number analyzed (Participants) | 221
participants | 9

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 9/221
Other Adverse Events (participants affected / at risk) | 0/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=221)
High LV Lead Threshold (Cardiac disorders) | 2 (2)
Infection (Surgical and medical procedures) | 2 (2)
LV Lead Dislodgement (Cardiac disorders) | 3 (3)
Lead Integrity Comprimised noted at Device Change-Out (Surgical and medical procedures) | 1 (1)
Phrenic Nerve Stimulation (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other